CLINICAL TRIAL: NCT02619357
Title: A Method Validation, Single-period, Open-label Evaluation Study to Explore the Sensitivity of a Novel Biosensor Device (SenseWear Armband Gecko) for Measuring Physical Activity in Subjects With COPD & Asthma
Brief Title: Method Validation Study to Explore the Sensitivity of SenseWear Armband Gecko for Measuring Physical Activity in Subjects With Chronic Obstructive Pulmonary Disease (COPD) & Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 202373
Record Dates: First submitted 2015-08-27; First posted 2015-12-02 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Asthma; wearable physical activity monitor; step counts; Exercise; energy expenditure; COPD; indirect calorimetry
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): 10 subjects diagnosed with COPD (GOLD stages 2 and 3). Subjects will wear multiple devices simultaneously (SenseWear Armband Gecko, SenseWear Armband MF, Actigraph GT9x wristband and waistband and Garmin Vivofit 2 wristband) up to 24 hours per day for 2 days while performing usual activities of daily living, strength exercises, laboratory-based, and field-based exercise tests.
  Interventions: Device: SenseWear Armband Gecko; Device: SenseWear Armband MF; Device: Actigraph GT9x wristband and waistband; Device: Garmin Vivofit 2 wristband; Device: SOMNOwatch plus EEG 6 sleep monitor; Other: Strength exercises; Other: Field-based exercise tests; Other: Laboratory-based exercise tests
- Cohort 2 (Experimental): 10 subjects diagnosed with asthma. Subjects will wear multiple devices simultaneously (SenseWear Armband Gecko, SenseWear Armband MF, Actigraph GT9x wristband and waistband and Garmin Vivofit 2 wristband) up to 24 hours per day for 2 days while performing usual activities of daily living, strength exercises, laboratory-based, and field-based exercise tests.
  Interventions: Device: SenseWear Armband Gecko; Device: SenseWear Armband MF; Device: Actigraph GT9x wristband and waistband; Device: Garmin Vivofit 2 wristband; Device: SOMNOwatch plus EEG 6 sleep monitor; Other: Strength exercises; Other: Field-based exercise tests; Other: Laboratory-based exercise tests

INTERVENTIONS:
Device: SenseWear Armband Gecko — Subjects will wear SenseWear Armband Gecko up to 24 hours per day for 2 days while performing usual activities of daily living, strength exercises, laboratory-based, and field-based exercise tests
Device: SenseWear Armband MF — Subjects will wear SenseWear Armband MF up to 24 hours per day for 2 days while performing usual activities of daily living, strength exercises, laboratory-based, and field-based exercise tests
Device: Actigraph GT9x wristband and waistband — Subjects will wear Actigraph GT9x wristband and waistband up to 24 hours per day for 2 days while performing usual activities of daily living, strength exercises, laboratory-based, and field-based exercise tests
Device: Garmin Vivofit 2 wristband — Subjects will wear Garmin Vivofit 2 wristband up to 24 hours per day for 2 days while performing usual activities of daily living, strength exercises, laboratory-based, and field-based exercise tests
Device: SOMNOwatch plus EEG 6 sleep monitor — In a subset of subjects, this device will be worn as a comparator for monitoring sleep quality and duration.
Other: Strength exercises — Subjects will perform strength exercises using elastic bands of varying resistance
Other: Field-based exercise tests — Subjects will perform an Incremental Shuttle Walk Test (ISWT) and each individual component of a Short Physical Performance Battery (SPPB).
Other: Laboratory-based exercise tests — Subjects will perform an incremental, symptom-limited cardiopulmonary exercise test on a cycle ergometer and will walk at various speeds on a treadmill

SUMMARY:
The prevalence, low cost, and low burden of wearable devices that provide quantitative and qualitative feedback on a subject's activity level present an opportunity for the use of these devices in clinical and observational studies. However, the accuracy and reproducibility of any given device may vary with device design and algorithm implementation. Therefore, validation of emerging technologies against known standards such as analysis of exhaled breath and currently available medical devices is critical. This is a single center, two-cohort, single period, open-label, methodology study. No investigational product will be used in this study. Eligible subjects will wear 2 generations of SenseWear Armband devices, 2 ActiGraph GT9x devices (one on the wrist and one on the waist) and a Garmin Vivofit 2 activity tracker wristband for up to 24 hours per day. Subjects who consent to participate in an optional sub-study will wear a SOMNOwatch Plus EEG-6 device while sleeping. Subjects will perform a variety of laboratory and field-based exercise tests and strength exercises using Latex-Free Therabands.The co-primary objectives of this study are firstly to compare the outputs of the test devices (SenseWear Armband Gecko and Actigraph GT9x) to those of the SenseWear Armband MF and secondly to assess the sensitivity and accuracy of the test devices in subjects with COPD or asthma while performing laboratory-based exercise testing.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1 (COPD) >=45 years and <=70 years
* Cohort 2 (Asthma) >=18 years and <=70 years.
* Cohort 1; subjects with a confirmed diagnosis of COPD (Gold stage 2 and 3, COPD patients will be classified according to Global Initiative for Chronic Obstructive Lung Disease [GOLD] Guidelines) as defined by post-bronchodilator spirometry FEV1 >=40% and <80% predicted, and FEV1/FVC <0.7
* Cohort 2; subjects with documented, physician-diagnosed asthma.
* BMI within the range 19 to 32 kilogram(kg)/m^2 (inclusive)
* Male or female; A female of childbearing potential is eligible to enter and participate in the study if she has a negative pregnancy test at screening and day 1.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* Women who are pregnant or lactating or are planning on becoming pregnant during the study.
* Alpha1-antitrypsin deficiency: Subjects with a diagnosis of alpha1-antitrypsin deficiency as the underlying cause of COPD, if known.
* Other respiratory disorders: Subjects with tuberculosis, lung cancer, significant bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung diseases or other active pulmonary diseases.
* Pneumonia or other respiratory tract infection that has not resolved at least 14 days prior to screening. In addition, any subject that experiences pneumonia during any period between the screening visit and the study visit will be excluded.
* COPD or asthma exacerbation (in this case defined as a change in symptoms requiring increased doses of current medicines or the prescription of new medicines, e.g., corticosteroids or antibiotics) that has not resolved at least 28 days prior to screening. COPD or asthma exacerbation during any period between the screening visit and the study visit will be excluded.
* Presence of severe and/or poorly controlled asthma that in the opinion of the investigator renders participation in the study unsafe
* Any co-morbid medical condition that in the opinion of the investigator would make participation in the study unsafe or unfeasible, including conditions that prohibit completion of exercise testing: orthopaedic, neurological, cardiovascular or other complaints that significantly impair normal biomechanical movement patterns and limit the ability to walk/cycle as judged by the investigator.
* Resting oxyhemoglobin saturation <94%.
* Use of supplemental oxygen therapy during the day or night.
* Drug/alcohol abuse: Subjects with a known or suspected history of alcohol (males >21 units per week and females >14 units per week) or drug abuse within the last 2 years. One unit is equivalent to 8 gram (g) of alcohol: a half-pint (~240 milliliter [mL]) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Inability to abstain from smoking during the period in which the subject is admitted to the Clinical Unit.
* A history of allergy or hypersensitivity to metal, particularly stainless steel.
* Clinically significant abnormality on electrocardiogram (ECG) as determined by the investigator.
* Any vital sign indicator, e.g., hypertension or tachycardia at rest that at the discretion of the investigator would make participation in the study unsafe or unfeasible.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-09-21 (Actual); Primary Completion 2016-03-16 (Actual); Study Completion 2016-03-16 (Actual)

PRIMARY OUTCOMES:
Energy expenditure [kilocalories per minute] | Up to Day 2
  Energy expenditure will be assessed by test devices at various levels of exertion during field-based and laboratory-based exercise tests. Graphical and/or statistical comparisons will be made between test devices and with information derived from indirect calorimetry obtained by exhaled gas analysis, where available.
Energy expenditure [metabolic equivalents] | Up to Day 2
  Energy expenditure will be assessed by test devices at various levels of exertion during field-based and laboratory-based exercise tests. Graphical and/or statistical comparisons will be made between test devices and with information derived from indirect calorimetry obtained by exhaled gas analysis, where available.
Step counts [total number of steps taken] | Up to Day 2
  Step counts will be collected by test devices at various levels of exertion during field-based and laboratory-based exercise tests. Graphical and/or statistical comparisons will be made between devices and with manually counted steps, where available.

SECONDARY OUTCOMES:
Number of subjects with adverse events (AE) or serious adverse events (SAE). | From the start of Study procedures until follow-up (6 days)
  AEs and SAEs will be collected for each subject from the start of study until the follow-up contact
Number of subjects with abnormal vital signs related to interventions. | Screening and Days 1 and 2
  Oral temperature (degrees Celsius), systolic and diastolic blood pressure (mmHg), heart rate (beats per minute), respiratory rate (breaths per minute), and oxygen saturation (percent) will be collected at various times throughout the study.
Forced Expiratory Volume in 1 second (FEV1) | Screening
  Post-salbutamol spirometry will be obtained at screening, if necessary. Post- salbutamol FEV1 will be determined.
Ratio of FEV1 and Forced Vital Capacity (FVC) | Screening
  Ratio of FEV1 and Forced Vital Capacity (FVC) will be determined at screening.
Borg dyspnea index score | Days 1 and 2
  Borg dyspnea scores will be obtained during and after exercise.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

REFERENCES:
- See also: Results for study 202373 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/202373?search=study&search_terms=202373#rs